CLINICAL TRIAL: NCT04079439
Title: Physical Activity With Tailored E-health Support for Individuals With Intellectual Disability (PA-IDe Study): a Randomised Controlled Trial
Brief Title: Physical Activity With Tailored E-health Support for Individuals With Intellectual Disability
Acronym: PA-IDe
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of COVID-19 the study was stopped. It has been changed to include a pilot trial, which has been conducted in 2021/2022 (trial registration: NCT04929106). The RCT will hopefully be conducted in the near future.
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HNF1353-17
Record Dates: First submitted 2019-08-20; First posted 2019-09-06 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2021-06

CONDITIONS: Intellectual Disability
MeSH Terms: conditions — Intellectual Disability | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two-armed randomised controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Tailored e-heath support for physical activity with a focus on communication and rewards, using commercial accelerometers for measurements
  Interventions: Behavioral: Physical activity with tailored e-health support
- Control group (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Physical activity with tailored e-health support — The planned e-health intervention will contain several elements: A motivating smartphone app registers indoor- and outdoor activity as well as activity from the use of an ergometer-bike. For recording of outdoor activity commercial wrist-born accelerometers will be used. The app-solution will be motivating and result in a reward after a predefined level of activity.
  Other Names: Activity planner
  Arms: Intervention

SUMMARY:
The main objective of this project is to enhance physical activity in youths and adults with intellectual disabilities (IDs) by developing and testing a tailored e-heath support for motivation and participation in physical activity.

DETAILED DESCRIPTION:
Individuals with intellectual disability (ID) have lower levels of physical activity and greater barriers for participation in fitness activities, compared to the general population. As increased physical activity has positive effects on cardiovascular and psychosocial health, identifying effective interventions for use in everyday settings is exceedingly important. E-health like motion sensor games (exergames) and smartphone reminders for physical activity have been explored and found to be promising in people with ID.

The purpose of this study is to examine the effectiveness of an individually tailored PA programme with motivational mobile e-health support on everyday level of PA in youths and adults with ID.

The PA-IDE trial uses a prospective randomized controlled design. In total, 60 participants with a sedentary lifestyle or low physical activity level will be included, aging from 16-60 years old. The intervention consists of a tailored e-health support intervention, using smartphones or tablets to create structure and predictability of physical activities. The intervention emphasizes the communicative abilities of individual participants and use rewards and give feedback of progress to motivate individuals to increase participation in physical activity. Participants will be allocated to groups consisting of 30 participants who receive either the e-health intervention or standard care (control). All participants will be assessed at baseline, 3-, and 6 months. Participants in the intervention group, close relatives or care staff will be invited to participate in a goal-setting meeting about physical activity in the intervention period, where the Goal Attainment Scaling (GAS) will be used. Primary outcome will be physical activity level measured as steps per day with commercial wrist-worn accelerometers. Secondary outcome measures include minutes of moderate activity, energy expenditure, social support for physical activity, self-efficacy in a PA setting, behaviour problems, and goal attainment.

The investigators expect that the new intervention will perform better than standard care in terms of improved physical activity, mastery, and social support for activities. Technology offers new opportunities to influence healthy behaviours. The trial results will determine the effectiveness and sustainability of a tailored e-health support intervention to increase physical activity among youths and adults with ID.

ELIGIBILITY:
Inclusion Criteria:

* Intellectual disability
* Age 15-60 years
* Low physical activity
* Sedentary lifestyle

Exclusion Criteria:

* Medical contradictions for participation
* High levels of physical activity

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Steps per day | Baseline, 3 months and 6 months
  The primary outcome is physical activity, objectively assessed by steps per day measured with an accelerometer. This will objectively assess physical activity and sedentary time. Change in steps per day is being assessed at baseline, after three months of intervention and after 6 months of intervention.

SECONDARY OUTCOMES:
Physical activity | Baseline, 3 months and 6 months
  The International Physical Activity Questionnaire - Short Form, adapted to measure PA using proxy respondents (IPAQ-SF) will be used. The IPAQ-SF is a 7-item questionnaire that assesses PA the last seven days at four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting.
Blood pressure | Baseline, 3 months and 6 months
  The blood pressure will be measured in units of millimeters of mercury (mmHg) using Welsh-Allyn device. Both systolic blood pressure and diastolic blood pressure will be measured.
Waist Circumference | Baseline, 3 months and 6 months
  Waist circumference will be measured in cm. Measurements will be done 1 cm above the navel.
Body Mass Index (BMI) | Baseline, 3 months and 6 months
  Height will be measured with a stadiometer (Seca) in meters, with the participant wearing no shoes. Weight measured with an analog, floor scale (Seca) in kilograms, with participants wearing no shoes or outdoors jacket/gears. For participants in wheelchair or with difficulty standing on a small plate a wheelchair weight (Seca) will be used. Weight and height will be combined to report BMI in kg/m^2.
Physical functioning | Baseline, 3 months and 6 months
  The Short Physical Performance Battery (SPPB) will used to assess physical functioning. The SPPB is a screening test designed to assess physical performance and predict disability in older population. The SPPB is mainly a measure of lower-extremity function and consists of three subtests; 1) Static balance: Standing balance is tested with the feet in the side-by-side, semi tandem and tandem positions for 10 s each; 2) Gait speed: a 4 meter (13ft) walk at the individual´s habitual pace.; 3) Lower limb strength as indicated by the ability to rise from a chair with folded arms across their chest.
Self-efficacy and social support | Baseline, 3 months and 6 months
  The Self-Efficacy/Social Support scales for Activity for persons with Intellectual Disability (SE/SS-AID) is a questionnaire consisting of four scales, where one scale measure self-efficacy for overcoming barriers to leisure PA. The last three scales measure social support for leisure activity from family members, residential staff, and friends with ID. The scale is validated for self-reporting from individuals with mild to moderate intellectual disability or can be used by proxy respondents. The questionnaire will be translated into the Norwegian language using standard guidelines.
Challenging behaviour | Baseline, 3 months and 6 months
  The Aberrant Behavior Checklist-Community (ABC-C) is a questionnaire designed to assess challenging behavior in children, youths and adults with an intellectual disability. The ABC is a 58-item checklist grouped into five subscales. It is a proxy measure requiring knowledge of the index person. Assigned weighted scores 0-3 (3 indicating most severe), grouped into five symptom-clusters (irritability, lethargy, stereotypy, hyperactivity, and inappropriate speech). The questionnaire has been validated for use in a Norwegian population with neurodevelopmental disabilities.
Satisfaction with life | Baseline, 3 months and 6 months
  Satisfaction of life is a scale developed by Bergström, Hochwälder, Kottorp, and Elinder (2013) for assessing satisfaction with home environment and leisure time among individuals with mild to moderate ID. The outcome is measured by four factors: 1) satisfaction with housing environment; 2) satisfaction with life; 3) satisfaction with meals; and 4) satisfaction with recreational activities. Items are read out load by a researcher and answered by 'good' (happy face = 2), 'in between' (neutral face = 1) and 'bad' (sad face = 0). In the current study the scale is used to control for adverse effects.
Social network | Baseline, 3 months and 6 months
  The Social Support scales for Activity for persons with Intellectual Disability (SS-AID) is a 17-item scale for measuring social support from family, paid staff and roommates with disabilities. The scale is self-report and validated for individuals with mild to moderate intellectual disability.
Goalsetting | Baseline, 3 months and 6 months
  The Goal attainment scale (GAS) will be used to identify self-management goals that participants want to achieve. The questionnaire will be filled out by the researcher, with participants and proxy respondents present. Completing the GAS involves several steps. Goals are selected by each individual and observable behavior that reflects a degree of goal attainment is defined. The participant's pre-treatment or baseline levels is defined in respect to the goal. Five different goal attainment levels are defined, ranging from "no change" to "much better than expected outcome" (numbered -2 to +2). Follow-up times for participant evaluation are set (presumably after 3- and 6 months). Participants are evaluated after the defined time interval. At the end, the overall attainment score for all goals are calculated. In this study we will define up to three goals for PA.

CONTACTS AND LOCATIONS:
Overall Officials: Audny Anke, Professor, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: Yes
A study protocol article will be published
Supporting Information: Study Protocol
Time Frame: The study protocol will be sent in and published during the year 2020.
Access Criteria: Study protocol will be published and will be available from publication date and forward.

REFERENCES:
- [Derived] Michalsen H, Wangberg SC, Hartvigsen G, Jaccheri L, Muzny M, Henriksen A, Olsen MI, Thrane G, Jahnsen RB, Pettersen G, Arntzen C, Anke A. Physical Activity With Tailored mHealth Support for Individuals With Intellectual Disabilities: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Jun 29;9(6):e19213. doi: 10.2196/19213. PMID 32437328